CLINICAL TRIAL: NCT02837133
Title: Effects of a Single Session of Integrated Yoga Therapy Compared With Other Relaxation Techniques
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hiroshima University (Other)
Responsible Party: Principal Investigator, Hitoshi Okamura, Professor, Institute of Biomedical & Health Sciences, Hiroshima University
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: HiroshimaU
Record Dates: First submitted 2016-07-07; First posted 2016-07-19 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Yoga

ARMS (1):
- other techniques group (Experimental): theory and practice of pair massage with tapping, stretching of the ankle and neck, and autogenic training
  Interventions: Behavioral: integrated yoga program

INTERVENTIONS:
Behavioral: integrated yoga program — the program as a one-time session for 3 hours as a component of a Stress Management Education program

SUMMARY:
Typically a course of yoga therapy for stress management takes place over a week, however, investigators are often asked to provide a single session for workers. The aim of this study is to assess the benefits of a single session of an integrated yoga program compared with other relaxation techniques for the staff of schools.

ELIGIBILITY:
Inclusion Criteria:

* school staff members, including school managers, teachers, school nurses, school office workers, nutritionists and cooks
* volunteers attending a stress management workshop

Exclusion Criteria:

* those who had any previous experience of practicing yoga or any relaxation procedures

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change of scores on the Subjective Units of Distress (SUD) scale | 1) immediately after the subjects arrived at the facility (baseline) and 2) immediately after the intervention
  SUD is a scale of 0 (comfort) to 10 (discomfort) for measuring the subjective intensity of disturbance or distress currently experienced by an individual covering both physical and mental aspects.